CLINICAL TRIAL: NCT03690882
Title: Medical Imaging Characteristics of Patient With Unclassified Acute Cervical Pain
Acronym: RetroTIPIC
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: CE_20151117_21_ALR
Record Dates: First submitted 2018-09-26; First posted 2018-10-01 (Actual); Last update posted 2018-10-01 (Actual); Status verified 2018-09

CONDITIONS: Carotidynia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cases of unclassified acute cervical pain
  Interventions: Other: systematic review of medical imaging

INTERVENTIONS:
Other: systematic review of medical imaging

SUMMARY:
Some cases of acute antero-lateral cervical pain cannot be accurately classified by medical imaging (ultrasound and/or magnetic resonance imaging and/or CT-scan) : imaging rules out carotid dissection, carotid occlusion or vasculitis as well as musculoskeletal causes and thus the pain is considered "of unknown origin".

The investigators hypothesize that in such cases perivascular inflammation of the carotid may be involved.

This study aims at systematically reviewing medical files (including imaging) of patients suffering from acute cervical pain in which carotid dissection, carotid occlusion or vasculitis as well as musculoskeletal causes have been ruled out by ultrasound and/or magnetic resonance imaging and/or CT-scan

ELIGIBILITY:
Inclusion Criteria:

* Adult patient with acute cervical pain
* Presence of at least one medical imaging modality of the neck : ultrasound with doppler imaging, magnetic resonance imaging, CT-scan
* Medical imaging of the neck includes dedicated vessel analysis
* Absence of definite diagnosis for the cause of the pain after imaging

Exclusion Criteria:

* Musculoskeletal cause of the pain
* Carotid dissection
* Carotid occlusion
* Carotid vasculitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients from 10 centers in France, who presented from January 2009 through April 2016 with acute cervical pain and with at least 1 diagnostic image (MR imaging, CT, or US including a dedicated vessel analysis) in which no clearly identified and classified vascular or musculoskeletal cause of the pain was found.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2016-03-01 (Actual)

PRIMARY OUTCOMES:
Proportion of cases with perivascular inflammation of the carotid on medical imaging | Within 2 weeks after the first consultation for acute cervical pain

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmologique A. de Rotchschild, Paris, France

IPD SHARING:
Plan to Share IPD: No